CLINICAL TRIAL: NCT06180876
Title: Effect of General Anesthesia With Remimazolam Versus Propofol on Postoperative Delirium in Elderly Patients
Brief Title: Effect of Remimazolam on Postoperative Delirium
Acronym: RED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJH-A-20220628
Record Dates: First submitted 2022-06-28; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: General Anesthetic Drug Adverse Reaction
Keywords: general anesthesia; elderly patients; remimazolam; propofol
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remimazolam (Experimental): remimazolam continuous infusion is used for general anesthesia; dosage:0.7-1.5mg/kg/h; duration: from start of anesthesia induction to end of surgery
  Interventions: Drug: remimazolam
- propofol (Active Comparator): propofol continuous infusion is used for general anesthesia; dosage:4-8mg/kg/h; duration: from start of anesthesia induction to end of surgery
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: remimazolam — continuous infusion
  Arms: remimazolam
Drug: propofol — continuous infusion
  Arms: propofol

SUMMARY:
Remimazolam is a novel benzodiazepine with ultra-short onset and offset of its effect. It can be used for general anesthesia. However, classical benzodiazepine such as midazolam was reported to increase the risk of postoperative delirium. Thus, the investigators aim to investigate the effect of remimazolam general anesthesia on postoperative delirium in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* patients scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* American Society of Anesthesiologists status ≥Ⅳ
* history of neurologic or psychiatric diseases
* difficulty in communication
* abuse of drug or alcohol
* suspected allergy to propofol or benzodiazepines

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-01-25 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
incidence of delirium by 3 days after surgery | from end of surgery to 3 days after surgery, in a total of 3 days

SECONDARY OUTCOMES:
incidence of delirium by 30 minutes after extubation | from extubation of tracheal tube to 30 minutes after extubation, in a total of 30 minutes
incidence of delirium by 1 day after surgery | from end of surgery to 1 day after surgery, in a total of 1 day
incidence of in-hospital delirium after surgery | from end of surgery to discharge from hospital, in an average of 5 days
time to awake | from end of surgery to response to verbal command, in an average of 10 minutes
incidence of hypotension during surgery | from start of anesthesia induction to extubation, in an average of 2 hours
  hypotension is defined as systolic blood pressure decreasing by more than 20% of baseline value
incidence of hypertension during surgery | from start of anesthesia induction to extubation, in an average of 2 hours
  hypertension is defined as systolic blood pressure increasing by more than 20% of baseline value
level of tumor necrosis factor α at the end of the surgery | at the end of the surgery
level of serum S100β at the end of the surgery | at the end of the surgery
level of interleukin α at the end of the surgery | at the end of the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Fourth military medical university, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Tang F, Yi JM, Gong HY, Lu ZY, Chen J, Fang B, Chen C, Liu ZY. Remimazolam benzenesulfonate anesthesia effectiveness in cardiac surgery patients under general anesthesia. World J Clin Cases. 2021 Dec 6;9(34):10595-10603. doi: 10.12998/wjcc.v9.i34.10595. PMID 35004991
- [Background] Liu T, Lai T, Chen J, Lu Y, He F, Chen Y, Xie Y. Effect of remimazolam induction on hemodynamics in patients undergoing valve replacement surgery: A randomized, double-blind, controlled trial. Pharmacol Res Perspect. 2021 Oct;9(5):e00851. doi: 10.1002/prp2.851. PMID 34390228
- [Background] Kilpatrick GJ. Remimazolam: Non-Clinical and Clinical Profile of a New Sedative/Anesthetic Agent. Front Pharmacol. 2021 Jul 20;12:690875. doi: 10.3389/fphar.2021.690875. eCollection 2021. PMID 34354587
- [Background] Doi M, Morita K, Takeda J, Sakamoto A, Yamakage M, Suzuki T. Efficacy and safety of remimazolam versus propofol for general anesthesia: a multicenter, single-blind, randomized, parallel-group, phase IIb/III trial. J Anesth. 2020 Aug;34(4):543-553. doi: 10.1007/s00540-020-02788-6. Epub 2020 May 16. PMID 32417976
- [Background] Oka S, Satomi H, Sekino R, Taguchi K, Kajiwara M, Oi Y, Kobayashi R. Sedation outcomes for remimazolam, a new benzodiazepine. J Oral Sci. 2021 Jun 29;63(3):209-211. doi: 10.2334/josnusd.21-0051. Epub 2021 Jun 7. PMID 34092775